

## **Assent Script**

# Parent Emotion Socialization and Child Emotion Regulation in FASD Principal Investigator: Christie L. M. Petrenko, Ph.D.

We are doing a research study.

## These are some things we want you to know about research studies:

Your parent or guardian needs to give permission for you to be in this study.

You do not have to be in this study if you don't want to, even if your parent has already given permission. If you start, you can stop being in the study at any time. No one will be mad if you want to stop.

## What will happen during this study?

We want to learn how kids think and feel.

If you take part, we will ask you to do things like:

- Play games on the computer
- Define words and solve problems
- Answer questions about your feelings
- Wear a special monitor to measure your heart rate
- Talk with your parent or guardian about things you've done as a family

We will meet with you three times. Once now, once in 3 months, and once 3 months after that. The first two times will last about 2 hours. The last time will be shorter and your part will only take 15 minutes.

## Who will be told the things we learn about you in this study?

The information we collect about you will be kept private. Only the people working on this study will be able to look at the information we collect. We will not tell anyone else anything you tell us unless we are worried about you or someone else.

## Will you get any money or gifts for being in this study?

You will receive money or a toy for being in this study. You will earn \$20 or a toy for the first two visits. On the third shorter visit, you will get to pick a small toy from a prize box.

Remember, being in this study is up to you and your parents. If you don't want to do this right now, just tell us. Even if your parent says you can be in this study, you don't have to.

If you start, you may stop at any time. If you decide to stop, no one will be mad at you.

187 Edinburgh Street · Rochester, NY 14608 585.275.2991 · 585.454.2972 *fax* 

RSRB Approval Date: 9/18/2020

| It is important that you understand what you will do in this study. Please ask us any questions you have. |
|---|
| What questions do you have? |
| Do you want to be in the study? |
| Subject Name: |
| (PRINTED BY Person Obtaining Assent) |
| Person Obtaining Assent I have read this form to the subject and/or the subject has read this form. An explanation of the research was given and questions from the subject were solicited and answered to the subject's satisfaction. In my judgment, the child has demonstrated comprehension of the information. I have given the child adequate time to consider the study before providing assent. My signature below documents the subject's assent to participate in this research study. |
| Name and Title (Print) |
| Signature of Person Obtaining Assent Date |

RSRB case number: 00069545 Page 2 of 2 Version Date: 7/30/2018